CLINICAL TRIAL: NCT06571227
Title: Establishing the Clinical Significance Values of the Lysholm Knee Score in Patients Undergoing Anterior Cruciate Ligament Reconstruction
Brief Title: Establishing the Clinical Significance Values of the Lysholm Knee Score
Status: Recruiting | Type: Observational
Sponsor: Kırklareli University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Ozan Gür, PT, Research Assistant, Kırklareli University
Other Study IDs: 2024 - 1202
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Knee Injuries
Keywords: Lsholm knee score; Anterior cruciate ligament injury; Minimal important change; Substantial clinical benefit; Clinical significance; Patient reported outcome
MeSH Terms: conditions — Knee Injuries; Anterior Cruciate Ligament Injuries | interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anterior Cruciate Ligament Reconstruction Patients: Patients who will undergo anterior cruciate ligament reconstruction because of anterior cruciate ligament rupture
  Interventions: Procedure: Anterior cruciate ligament reconstruction

INTERVENTIONS:
Procedure: Anterior cruciate ligament reconstruction — Patients with anterior cruciate ligament rupture will undergo anterior cruciate ligament reconstruction surgery.

SUMMARY:
The goal of this observational study is to learn about patients who will undergo anterior cruciate ligament reconstruction. The main questions it aims to answer are:

* What is the minimal clinically important difference value of the Lysholm Knee Score?
* What is the substantial clinical benefit value of the Lysholm Knee Score?
* What are the risk factors that prevent patients who have undergone anterior cruciate ligament reconstruction from reaching the minimal clinically important difference value?
* What are the risk factors that prevent patients who have undergone anterior cruciate ligament reconstruction from reaching the substantial clinical benefit value?

ELIGIBILITY:
Inclusion Criteria:

* to be over 18 years old
* to undergo surgery for a ruptured anterior cruciate ligament

Exclusion Criteria:

* to have metabolic or autoimmune diseases
* to undergo revision anterior cruciate ligament surgery or anterior cruciate ligament repair
* to have cognitive issues that will hinder the completion of the study forms
* to lack sufficient proficiency in Turkish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted with people undergoing anterior cruciate ligament reconstruction at Gazi University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Functional level | before the surgery and after 3 months from the surgery
  Lysholm Knee Score (total score between 0-100) (higher values indicate higher functional level)

CONTACTS AND LOCATIONS:
Overall Officials: Ozan Gür, MSc, Principal Investigator — Kırklareli University
Locations (1):
- Gazi Üniversitesi Hastanesi, Ankara, Turkey (Türkiye)